CLINICAL TRIAL: NCT04236856
Title: An Evaluation of Effectiveness and Safety of the CorPath® GRX System in Endovascular Embolization Procedures of Cerebral Aneurysms
Brief Title: CorPath® GRX Neuro Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-08660
Record Dates: First submitted 2020-01-02; First posted 2020-01-22 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage; Headache
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Headache

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, international, multi- center, non-inferiority study to evaluate the effectiveness and safety of the CorPath GRX System for endovascular cerebral aneurysm embolization compared to historical controls.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic Endovascular Procedure (Other): Subjects with a clinical indication for endovascular coil and/or stent assisted coiling embolization of cerebral aneurysms will be treated using the CorPath GRX System.
  Interventions: Device: Robotic Endovascular Procedure

INTERVENTIONS:
Device: Robotic Endovascular Procedure — After providing written informed consent, subjects with cerebral aneurysms may have their aneurysm treated using the CorPath GRX System.
  Other Names: CorPath GRX System

SUMMARY:
The primary objective of this study is to evaluate the effectiveness and safety of robotic-assisted endovascular embolization procedures compared to objective performance criteria for traditional, manual operation based on the scientific literature.

DETAILED DESCRIPTION:
This is a prospective, single-arm, international, multi- center, non-inferiority study to evaluate the effectiveness and safety of the CorPath GRX System for endovascular cerebral aneurysm embolization compared to historical controls. Subject selection requires a clinical indication for endovascular coil and/or stent-assist coiling embolization of cerebral aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. At least one cerebral aneurysm (unruptured) with indication for endovascular treatment; dome to neck ratio >1.5 or aneurysm neck width >4.0 mm.
3. The Investigator deems the procedure appropriate for both manual or robotic-assisted endovascular treatment.
4. The conscious subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Failure / unwillingness of the subject to provide informed consent, unless the EC has waived informed consent.
2. The Investigator determines that the subject or the neurovascular anatomy is not suitable for robotic-assisted endovascular treatment.
3. Women who are pregnant.
4. Persons under guardianship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-04-23 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Piotin, MD, PhD, Principal Investigator — Interventional Neuroradiologisit & Director, Foundation Rothschild
Locations (10):
- Gold Coast University Hospital, Southport, Queensland, Australia
- Uniklinikum Salzburg, Salzburg, Austria
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto
- France (3):
  - Hôpital Pitié-Salpêtrière, Paris, CA
  - CHU Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Hôpital de la Fondation Rothschild, Paris
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona
  - University Clinical Hospital of Valladolid, Valladolid
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD.

REFERENCES:
- [Background] Lawton MT, Vates GE. Subarachnoid Hemorrhage. N Engl J Med. 2017 Jul 20;377(3):257-266. doi: 10.1056/NEJMcp1605827. No abstract available. PMID 28723321
- [Background] Lantigua H, Ortega-Gutierrez S, Schmidt JM, Lee K, Badjatia N, Agarwal S, Claassen J, Connolly ES, Mayer SA. Subarachnoid hemorrhage: who dies, and why? Crit Care. 2015 Aug 31;19(1):309. doi: 10.1186/s13054-015-1036-0. PMID 26330064
- [Background] Connolly ES Jr, Rabinstein AA, Carhuapoma JR, Derdeyn CP, Dion J, Higashida RT, Hoh BL, Kirkness CJ, Naidech AM, Ogilvy CS, Patel AB, Thompson BG, Vespa P; American Heart Association Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular Nursing; Council on Cardiovascular Surgery and Anesthesia; Council on Clinical Cardiology. Guidelines for the management of aneurysmal subarachnoid hemorrhage: a guideline for healthcare professionals from the American Heart Association/american Stroke Association. Stroke. 2012 Jun;43(6):1711-37. doi: 10.1161/STR.0b013e3182587839. Epub 2012 May 3. PMID 22556195
- [Background] Steiner T, Juvela S, Unterberg A, Jung C, Forsting M, Rinkel G; European Stroke Organization. European Stroke Organization guidelines for the management of intracranial aneurysms and subarachnoid haemorrhage. Cerebrovasc Dis. 2013;35(2):93-112. doi: 10.1159/000346087. Epub 2013 Feb 7. PMID 23406828
- [Background] Keedy A. An overview of intracranial aneurysms. Mcgill J Med. 2006 Jul;9(2):141-6. PMID 18523626
- [Derived] Mendes Pereira V, Rice H, De Villiers L, Sourour N, Clarencon F, Spears J, Tomasello A, Hernandez D, Cancelliere NM, Liu XYE, Nicholson P, Costalat V, Gascou G, Mordasini P, Gralla J, Martinez-Galdamez M, Galvan Fernandez J, Killer-Oberpfalzer M, Liebeskind DS, Turner RD, Blanc R, Piotin M. Evaluation of effectiveness and safety of the CorPath GRX robotic system in endovascular embolization procedures of cerebral aneurysms. J Neurointerv Surg. 2024 Mar 14;16(4):405-411. doi: 10.1136/jnis-2023-020161. PMID 37793795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation started with enrollment of first subject on 21 August 2020 and subject recruitment was completed on 21 April 2022. With 10 investigational sites, up to 120 subjects were enrolled in order to achieve at least 108 subjects in the study; each site was initially approved to recruit a maximum of 20 subjects. The total study duration was 24 months: the recruitment phase was 18 months and follow-up continues to 180 days.
Period: Overall Study
Arm/Group | Robotic Endovascular Procedure
Started | 120
Completed | 117
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 56.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 30
  Austria | 2
  France | 49
  Australia | 24
  Switzerland | 3
  Spain | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedural Technical Success.
Description: The primary effectiveness endpoint will be defined as successful completion of the robotic-assisted endovascular procedure absent any unplanned conversion to manual for guidewire or microcatheter navigation, embolization coil(s) or intracranial stent(s) deployment, or an inability to navigate vessel anatomy.
Time Frame: Measured from the start of the procedure to the end of the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
Participants | 110

2. Primary Outcome: Number of Intra- and Peri-procedural Events.
Description: The primary safety endpoint will be a composite of intra- and periprocedural events, including target aneurysmal rupture, vessel perforation or dissection, and thromboembolic event with neurological decline within 24-hours post- procedure or hospital discharge, whichever occurs first.
Time Frame: Measured from the start of the procedure through 24 hours or discharge, whichever occurs first.
Measure: Number; unit: Events
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
Events | 4

3. Secondary Outcome: Robotically Navigate Device to the Target Aneurysm
Description: Defined as successful advancement of device to the target aneurysm robotically.
Time Frame: Measured from the start of the procedure to the end of the procedure. Measured from the start of the procedure to the end of the procedure.
Reporting Status: Not Posted

4. Secondary Outcome: Robotically Deploy Therapeutic Device Into the Target Aneurysm
Description: Defined as successful deployment of therapeutic device into the target aneurysm robotically
Time Frame: as for outcome 3
Reporting Status: Not Posted

5. Secondary Outcome: Overall Procedure Time
Description: Defined as the time measured from the insertion of the access sheath/catheter until the removal of the microcatheter
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
minutes | 117.3 (47.3)

6. Secondary Outcome: Fluoroscopy Time
Description: Total fluoroscopy utilized during the procedure as recorded by the Imaging System
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
minutes | 51.9 (27.4)

7. Secondary Outcome: Patient Radiation Exposure
Description: DAP (dose-area-product) and/or AK (Air Kerma) as recorded during the procedure
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: mGy*cm2
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 104
mGy*cm2 | 6886135.5 (25767850.8)

8. Secondary Outcome: Contrast Fluid Volume
Description: Total contrast used during the procedure
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 116
cc | 185.4 (82.3)

9. Secondary Outcome: Adverse Events
Description: All adverse events (AEs) from the start of the CorPath GRX procedure until the end of the study will be summarized;
Time Frame: Measured from the start of the procedure through end of the study. Measured from the start of the procedure to the end of the procedure. Measured from the start of the procedure to the end of the procedure. Subjects will undergo clinical follow-up th
Reporting Status: Not Posted

10. Secondary Outcome: Number of Thromboembolic Events
Description: Rate of thromboembolic events occurring up to 180-days following the robotic-assisted procedure
Time Frame: Measured from the start of the procedure through end of the study (180-days following the robotic-assisted procedure).
Measure: Number; unit: Events
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 117
Events | 17

11. Secondary Outcome: Devices Used Robotically
Description: Recorded as successful or unsuccessful in conjunction with the CorPath GRX System
Time Frame: Measured from the start through end of the procedure. Subjects will also undergo clinical follow-up through 180 day
Reporting Status: Not Posted

12. Secondary Outcome: Number of Participants With Aneurysm Occlusion
Description: Angiographic assessment of aneurysm occlusion grade according to the Raymond-Roy Occlusion Classification Scale, parent-vessel compromise, and occlusion durability as assessed from an independent core laboratory.
  Raymond Roy Occlusion Classification Scale - Minimum:1, Maximum: 3b, Higher score meaning worse outcome.
Time Frame: Assessed at 180 Day Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 102
Participants
  Raymond Roy Classification Scale 1 | 96
  Raymond Roy Classification Scale 2 | 2
  Raymond Roy Classification Scale 3A | 2
  Raymond Roy Classification Scale 3B | 2

13. Secondary Outcome: Number of Participants With Aneurysm Occlusion
Description: as for outcome 12
Time Frame: Assessed During Procedure (Post Intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Endovascular Procedure
Number analyzed (Participants) | 110
Participants
  Raymond Roy Classification Scale 1 | 71
  Raymond Roy Classification Scale 2 | 5
  Raymond Roy Classification Scale 3A | 28
  Raymond Roy Classification Scale 3B | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Robotic Endovascular Procedure
All-Cause Mortality (participants affected / at risk) | 1/117
Serious Adverse Events (participants affected / at risk) | 40/117
Other Adverse Events (participants affected / at risk) | 21/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic Endovascular Procedure (N=117)
Stroke (Nervous system disorders) | 17
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 4
Transient Ischemic Attack (Nervous system disorders) | 3
Aphasia (Nervous system disorders) | 1
Confusion Episode (Nervous system disorders) | 1
Digestive Bleeding (Gastrointestinal disorders) | 1
Embolism (Blood and lymphatic system disorders) | 1
Extremity Ischemia (Vascular disorders) | 1
Fibula Fracture (Musculoskeletal and connective tissue disorders) | 1
Flow Diverter Endovascular Procedure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Intraprocedural Aneurysm Rupture (Nervous system disorders) | 2
Perforated Sigmoid Diverticulitis (Injury, poisoning and procedural complications) | 1
Relapsed Leukemia (Blood and lymphatic system disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Revascularization (Nervous system disorders) | 1
Right radial pseudoaneurysm (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Robotic Endovascular Procedure (N=117)
Headache (Nervous system disorders) | 8
Vascular Site Access Complication (Injury, poisoning and procedural complications) | 2
Electrolyte Disorder (Endocrine disorders) | 2
Confusion Episode (Nervous system disorders) | 1
Sensory Deficit (Nervous system disorders) | 1
Tinnitus (Nervous system disorders) | 2
Diabetes (Endocrine disorders) | 1
Galactorrhea (Endocrine disorders) | 1
Hemianopia (Eye disorders) | 1
Urine Infection (Infections and infestations) | 1
Vasospasm (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT04236856/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT04236856/SAP_001.pdf